CLINICAL TRIAL: NCT00575822
Title: Endoscopic Full-Thickness Plication for the Treatment of Gastroesophageal Reflux Disease: A Randomized, Sham-Controlled Trial
Brief Title: A Study to Determine the Effectiveness of Endoscopic Full-Thickness Plication for the Treatment of GERD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsoring company ceased business operations.
Sponsor: NDO Surgical, Inc. (Industry)
Responsible Party: Bruce R. Gaumond, Associate Director, Clinical Affairs, NDO Surgical, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 135-01885
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2008-05

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: GERD; Sham; Randomized Controlled Study; Endoscopic Full-thickness Plication; Plicator
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): NDO Endoscopic Full-thickness Plicator procedure
  Interventions: Device: NDO Full-thickness Plicator
- 2 (Sham Comparator): Sham control procedure
  Interventions: Device: Sham Control

INTERVENTIONS:
Device: NDO Full-thickness Plicator — A low-profile (≤6mm) gastroscope was advanced and an EGD followed by Savary wire placement was performed. The gastroscope was then removed and the Plicator was advanced directly over the wire and into the stomach. The gastroscope was re-introduced through the Plicator, and the Plicator was retroflexed under direct endoscopic visualization to the anterior gastric cardia, approximately 1cm below the gastroesophageal (GE) junction. The Plicator arms were opened and the endoscopic tissue retractor was advanced deeply into the gastric cardia. The gastric wall was then retracted into the open arms of the Plicator. The arms were closed and a single, transmural pledgeted suture was deployed. The Plicator and gastroscope were then removed and the gastroscope re-inserted to evaluate the post-plication GE junction.
  Other Names: Active Plicator procedure
  Arms: 1
Device: Sham Control — The sham procedure was identical to the treatment procedure through the positioning of the retroflexed Plicator 1cm below the GE junction. The Plicator instrument remained in this position for 15 minutes, based on average procedure times established in previous studies. During the sham procedure, physician investigators were required to talk through the procedure steps to maintain the patient blind.
  Other Names: Sham control procedure
  Arms: 2

SUMMARY:
The aim of this study was to determine the effectiveness of endoscopic full-thickness plication (Plicator; NDO Surgical, Inc., Mansfield, MA) for the treatment of GERD in comparison to a sham procedure.

Patients with symptomatic GERD requiring maintenance proton pump inhibitor therapy were entered into a randomized, single-blind, prospective, multicenter trial. Seventy-eight patients were randomly assigned to undergo endoscopic full-thickness restructuring of the gastric cardia with transmural suture. Eighty-one patients underwent a sham procedure. Group assignments were revealed following the 3-month evaluation. The primary endpoint was ≥ 50% improvement in GERD-HRQL score. Secondary endpoints included medication use and esophageal acid exposure.

Patients achieving ≥ 50% improvement in GERD-HRQL score at 3-months versus baseline off-meds were considered responsive to their assigned procedure. Patients who failed to reach this level of improvement at 3-months were considered non-responders. Analysis of these dichotomized variables (responder/non-responder) was done using Fisher's exact test comparing the proportion of responders between the active and sham groups. Intent-to-treat analysis was also performed. The null hypothesis was that the proportion of responders was the same in both the active and sham groups. Testing was done at the 5% level of significance (alpha=0.05).

ELIGIBILITY:
Patients 18 years or older with a history of heartburn or regurgitation symptoms requiring daily PPI therapy were recruited.

Inclusion Criteria:

* GERD-HRQL score ≥ 15 while off PPI therapy, and at least 6 points higher than on-PPI score
* Pathologic esophageal acid exposure, defined as pH<4.0 ≥ 4.5% of a 24- or 48-hour monitoring period or a DeMeester score > 14.7
* Lower esophageal resting pressure of at least 5mmHg; and
* Suitability for surgery (American Society of Anesthesiologists Physical Status Classification I or II).

Exclusion Criteria:

* Significant esophageal dysmotility as determined by manometry
* Esophagitis grade III or IV (Savary-Miller)
* Barrett's epithelium
* Hiatus hernia > 2cm
* Persistent dysphagia, weight loss, esophageal bleeding, vomiting, gas or bloating
* Esophageal or gastric varices
* Previous endoscopic or surgical anti-reflux procedure
* Other esophageal or gastric surgery
* Chronic use of anticoagulant or platelet anti-aggregation therapy (other than for cardiac prophylaxis); and
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2005-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
>/=50% improvement in GERD-Health Related Quality of Life Score | 3-months post-procedure

SECONDARY OUTCOMES:
GERD medication use | 3-months post-procedure
Esophageal acid exposure | 3-months post-procedure
Heartburn score as measure by visual analog scale | 3-months post-procedure
Quality of Life as measure by SF-36 | 3-months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Richard Rothstein, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center, Lebanon, NH; Charles Filipi, MD, Principal Investigator — Creighton University Medical Center, Omaha, NE; Karel Caca, MD, Principal Investigator — Klinikum Ludwigsburg, University of Heidelburg, Heidelburg, Germany; Ronald Pruitt, MD, Principal Investigator — Nashville Medical Research and the Maria Nathanson Center of Excellence, Nashville, TN; Klaus Mergener, MD, Principal Investigator — Digestive Health Specialists, Tacoma, WA; Alfonso Torquati, MD, Principal Investigator — Vanderbilt University Medical Center, Nashville, TN; Gregory Haber, MD, Principal Investigator — Lenox Hill Hospital, New York, NY; Yang Chen, MD, Principal Investigator — University of Colorado Health Science Center, Denver, CO; Kenneth Chang, MD, Principal Investigator — University of California at Irvine Medical Center, Orange, CA; David Wong, MD, Principal Investigator — Tri Valley Gastroenterology, San Ramon, CA; Jacques Deviere, MD, Principal Investigator — Erasme Hospital, Brussels, Belgium; Douglas Pleskow, MD, Principal Investigator — Beth Israel Deaconess Medical Center, Boston MA; Charles Lightdale, MD, Principal Investigator — Columbia University Medical Center, New York, NY; Alain Ades, MD, Principal Investigator — Seacoast Gastroenterology, Exeter, NH; Richard Kozarek, MD, Principal Investigator — Virginia Mason Medical Center, Seattle, WA
Locations (15):
- United States (13):
  - University of California at Irvine Medical Center, Orange, California
  - Tri Valley Gastroenterology, San Ramon, California
  - University of Colorado Health Science Center, Denver, Colorado
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Creighton University Medical Center, Omaha, Nebraska
  - Seacoast Gastroenterology, Exeter, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Lenox Hill Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Nashville Medical Research and the Maria Nathanson Center of Excellence, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Virginia Mason Medical Center, Seattle, Washington
  - Digestive Health Specialists, Tacoma, Washington
- Erasme Hospital, Brussels, Belgium
- Klinikum Ludwigsburg, University of Heidelburg, Heidelberg, Germany

REFERENCES:
- [Result] Rothstein R, Filipi C, Caca K, Pruitt R, Mergener K, Torquati A, Haber G, Chen Y, Chang K, Wong D, Deviere J, Pleskow D, Lightdale C, Ades A, Kozarek R, Richards W, Lembo A. Endoscopic full-thickness plication for the treatment of gastroesophageal reflux disease: A randomized, sham-controlled trial. Gastroenterology. 2006 Sep;131(3):704-12. doi: 10.1053/j.gastro.2006.07.004. PMID 16952539